CLINICAL TRIAL: NCT07285018
Title: Randomized, Placebo-Controlled, Phase 2 Clinical Trial to Evaluate LY4065967 for the Treatment of Diabetic Peripheral Neuropathic Pain
Brief Title: A Chronic Pain Master Protocol (CPMP): A Study of LY4065967 in Participants With Diabetic Peripheral Neuropathic Pain
Acronym: NP07
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27370; H0P-MC-NP07 (Other: Eli Lilly and Company); H0P-MC-CPMP (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-12-09; First posted 2025-12-16 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Diabetic Peripheral Neuropathic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY4065967 (Experimental): Participants will receive LY4065967 orally.
  Interventions: Drug: LY4065967
- Placebo (Placebo Comparator): Participants will receive placebo orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY4065967 — Administered orally
  Arms: LY4065967
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the safety and efficacy of study drug LY4065967 for the treatment of diabetic peripheral neuropathic pain (DPNP). This trial is part of the chronic pain master protocol H0P-MC-CPMP (NCT05986292) which is a protocol to accelerate the development of new treatments for chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Have presence of diabetic peripheral neuropathy, of symmetrical nature and in lower extremities for ≥6 months and diagnosed by a score of Part B ≥3 on Michigan Neuropathy Screening Instrument (©University of Michigan)
* Have a history and current diagnosis of type 1 or type 2 diabetes mellitus.
* Have an HbA1c <11% and on a stable regimen for treatment of diabetes at least 90 days prior to screening
* Have a body mass index at screening of ≤40 kilogram per meter squared (kg/m2)

Exclusion Criteria:

* Are pregnant or breastfeeding
* Have a history of other potentially causative and/or confounding sources of pain that may impair self-assessment of pain due to diabetic peripheral neuropathic pain (DPNP)
* Have lower limb amputation due to diabetes inclusive of great toe (metatarsal bone)
* Have serum vitamin B12 ≤200 picogram per milliliter (pg/mL)
* Have an abnormal BP (systolic BP >140 mm Hg and diastolic BP>90 mm Hg) at screening
* Have history or current clinically significant cardiac disease, including arrhythmia, aortic aneurysm, heart failure, current electrolyte abnormalities, or any other conditions that could predispose to arrhythmia in the judgement of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Average Pain Intensity as Measured by the Numeric Rating Scale (NRS) | Baseline, Week 8

SECONDARY OUTCOMES:
Change From Baseline in the Brief Pain Inventory-Short Form Modified (BPI-SFM) Total Pain Interference Score | Baseline, Week 8
Change from Baseline in Overall Improvement as Measured by Patient's Global Impression of Change (PGI-C) | Baseline, Week 8
Change from Baseline in Worst Pain Intensity as Measured by NRS | Baseline, Week 8
Change from Baseline in Sleep Scale from the Medical Outcomes Study (MOS Sleep Scale) | Baseline, Week 8
Change from Baseline in Emotional Functioning as Measured by the EuroQol-5D 5 Level Questionnaire (EQ 5D 5L) | Baseline, Week 8
Total Amount of Rescue Medication Used Daily During the Treatment Phase | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (37):
- United States (36):
  - Central Research Associates, Birmingham, Alabama
  - Central Phoenix Medical Clinic, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Desert Oasis Healthcare Medical Group, Palm Springs, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - CMR of Greater New Haven, Hamden, Connecticut
  - Bradenton Research Center, Inc., Bradenton, Florida
  - Accel Research Sites - DeLand Clinical Research Unit, DeLand, Florida
  - K2 MEDICAL Research THE VILLAGES, Lady Lake, Florida
  - K2 Medical Research ORLANDO, Maitland, Florida
  - Merritt Island Medical Research, LLC, Merritt Island, Florida
  - Suncoast Research Group, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Renstar Medical Research, Ocala, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Charter Research - Lady Lake, The Villages, Florida
  - Conquest Research, Winter Park, Florida
  - North Georgia Clinical Research, Woodstock, Georgia
  - Northwestern University, Chicago, Illinois
  - DelRicht Research, New Orleans, Louisiana
  - Lucida Clinical Trials, New Bedford, Massachusetts
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Rochester Clinical Research, LLC, Rochester, New York
  - Lillestol Research, Fargo, North Dakota
  - META Medical Research Institute, Dayton, Ohio
  - DelRicht Research, Tulsa, Oklahoma
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - FutureSearch Trials of Neurology, Austin, Texas
  - Re:Cognition Health - Fort Worth, Fort Worth, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - Rainier Clinical Research Center, Renton, Washington
- Ponce Medical School Foundation Inc., Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/